CLINICAL TRIAL: NCT04877236
Title: Pilot Trial Green Sun Medical Dynamic Brace
Brief Title: Green Sun Medical Dynamic Brace
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No interest in pursuing study
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Kenneth Illingworth, Principal Investigator, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-19-00293
Record Dates: First submitted 2021-04-29; First posted 2021-05-07 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Adolescent Idiopathic Scoliosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Green Sun Medical Brace (Experimental): This study only has one arm, administration of the Green Sun Medical Whisper Brace.
  Interventions: Device: Green Sun Medical Brace

INTERVENTIONS:
Device: Green Sun Medical Brace — All patients in the study will receive the Green Sun Medical Whisper Brace. Each GSM brace will be custom-fabricated via computer-assisted design using the 3D torso scans and a treatment plan (e.g. placement of corrective forces) devised by the treating orthotist as inputs. The brace components are then assembled. Once fabricated, the GSM brace will be fit to the subject by representatives of the manufacturer and in consultation with the treating orthotist.
  The GSM brace will be prescribed for the same number of hours per day as was the TLSO (generally 18-22 hours per day, individualized based on patient characteristics). Subjects and the family will be shown how to don and doff the brace, how to clean the brace cover, how to remove the temperature monitor, and how to remove the iButton and how to replace batteries in the GSM sensor board.

SUMMARY:
The Green Sun Medical Dynamic Brace (GSM) brace was developed as an alternative to rigid thoracolumbosacral orthoses (TLSOs, braces) commonly used to prevent continued curve progression in patients with adolescent idiopathic scoliosis (AIS). The brace applies corrective forces to the muscular and bony structures of the spine while preserving range of motion (ROM). The innovative design of this brace should provide an equivalent degree of correction of the scoliotic curvature as a rigid TLSO, with increased acceptability to the patient via improved comfort and spinal/chest wall mobility. Increased acceptability promotes increased adherence to treatment. This is a pilot study to collect preliminary short-term data concerning the safety and performance of the GSM brace in a sample of subjects with AIS who are currently being treated with a TLSO. The study will use clinical exams, x-rays, monitoring equipment, and questionnaires to primarily assess safety and performance. Secondary endpoints include spinal ROM and lung vital capacity assessment, as well as data validation. The study involves 3 visits, a performance check phone call, and 4 follow up calls over a four month span. This is a pilot study and no formal hypothesis testing will be done. Descriptive statistics of selected variables will be calculated.

DETAILED DESCRIPTION:
The Green Sun Medical Dynamic Brace (GSM) brace was developed as an alternative to rigid thoracolumbosacral orthoses (TLSOs, braces) commonly used to prevent continued curve progression in patients with adolescent idiopathic scoliosis (AIS). The brace applies corrective forces to the muscular and bony structures of the spine while preserving range of motion (ROM). The orthosis is prefabricated and adjusted for each patient. A series of semi-rigid segments encircle the patient's torso in close contact and are joined by a structure of flexible elements. These flexible (or elastic) elements generate stabilizing forces, providing the necessary immobilization while allowing relative motion of the semi-rigid segments. To date, this brace has been tested in the lab on healthy volunteers.

The innovative design of this brace should provide an equivalent degree of correction of the scoliotic curvature as a rigid TLSO, with increased acceptability to the patient via improved comfort and spinal/chest wall mobility. Increased acceptability promotes increased adherence to treatment. Given the strong research evidence that bracing effectiveness is a function of correction and adherence, there is reason to believe that a future pivotal study of the GSM brace could demonstrate superior effectiveness to rigid TLSO designs.

This is a pilot study to collect preliminary short-term data concerning the safety and performance of the GSM brace in a sample of subjects with AIS who are currently being treated with a TLSO.

In addition, this pilot study to provide "proof of concept" data which will inform further refinements of the GSM brace and support the development of a subsequent pivotal multicenter clinical trial.

Our primary aims involve safety and performance.

This is a multi-center, open-label trial where subjects serve as their own controls. Baseline radiographic and patient report will reflect the effect of the subject's standard of care TSLO, providing data that can be directly compared to that obtained during use of the GSM brace.

Immediately After Consent is Signed and Received by Study Team

The following will be sent to Green Sun so that an appropriately-configured GSM can be made for the subject:

1. A de-identified copy of the most recent 3D scan of the patient's torso (tagged with a study ID number)
2. The individualized treatment plan devised by the PI which specifies the location and direction of applied forces (e.g. push on the patient's left axilla, push on the patient's right rib cage roughly 4 inches lateral of midline around T9) and tagged with a study ID number The Baseline Visit will be scheduled approximately 2 weeks after consent is signed and the 3D scan and treatment plan have been sent to Green Sun to allow Green Sun time to fabricate the brace.

Instructions for Radiographs

1. All study-related radiographs will be obtained using the EOS® Imaging system Micro Dose protocol as available. If not, Standard of Care measures can be employed
2. The number of study-related radiographs is NOT to exceed 6.
3. Three radiographs are required:

   1. In the TLSO (Baseline Visit 1)
   2. In the GSM (Visit 2)
   3. Out of brace (Visit 3)
4. A maximum of 3 optional in-brace radiographs may be taken at any time prior to Visit 3 to maximize the fit, correction and comfort of the GSM brace.

Baseline Visit 1 (approximately 2 hours)

1. A urine pregnancy test will be conducted. Pregnant subjects will exit the study.
2. Completion of the Brace Questionnaire and the Italian Spine Youth Quality of Life (ISYQOL) questionnaire (5 minutes)
3. Assessments while wearing current TLSO

   1. Vital capacity using Spiropet spirometer (average of 3 trials, 5 minutes)
   2. Measurement of spine range-of-motion (flexion, extension, rotation) using a tape measure (5 minutes)
   3. In-brace standing coronal full-spine radiograph (5 minutes)
4. The subject will be fitted with the customized GSM brace. The fit and corrective forces will be fine-tuned by adjusting the drive mechanisms until the corrective forces are matched to the surface anatomy of the patient and to the spinal deformity. The subject is involved in this process by providing feedback concerning the comfort of the brace and the brace cover. A log will be kept of all adjustments made to the brace during the course of the study. The brace will include the embedded force and acceleration sensors, as well as two temperature monitor (Orthotimer or iButton) units.
5. Assessments while wearing Green Sun Brace

   1. Vital capacity using Spiropet (average of 3 trials, 5 minutes)
   2. Measurement of spine range-of-motion (flexion, extension, rotation) using a tape measure (5 minutes)
6. Subject sent home with daily GSM Brace Diary
7. Extraction of data from medical/orthotic records: date of birth, gender, date of menses onset, and historical measures of height, weight, skeletal maturity (Risser grade, status of triradiate), Scoliosis Research Society curve classification, Cobb angle(s), kyphosis, lordosis, coronal and sagittal balance, apical vertebral rotation, in-brace Cobb angle(s) and estimated brace wear time. Data from TLSO brace initiation to baseline study visit will be extracted. These data define the spinal deformity, and the risk for continued progression.
8. OPTIONAL: Subject Appraisal of the GSM Brace Wear Mobile App Subjects will be given the option to use and provide feedback concerning the GSM mobile app (Dynamic Scoliosis Brace Monitoring App, Version 1.5.1, developed by Green Sun Medical and Mindset Medical). This app pairs the subject's mobile device with the GSM sensor in the brace and offloads date, accelerometer and pressure sensor data to estimate the number of hours per day that the brace is being worn by the patient. The app graphically displays the estimated hours/day the brace was worn for the current day and for the week. The app provides real-time feedback using graphical displays that should be easily understandable by adolescents. There is research evidence that providing subjects with brace wear time feedback results in better compliance to brace wear recommendations. 9, 16 Subjects will be given the option to use the app and to complete the GSM App feedback form at Visit 2 and Visit 3. The purpose of the app in this study is not to assess brace wear time or the influence of the app on wear time, but only to gather subjects' opinions for ongoing refinement of the app. The accuracy or reliability of the app is not being tested in this study. Subject PHI will not be used for registration; subjects will be instructed to enter their Study ID and City instead of their First and Last names; DOB as January 1, 2019; their email will be entered as the StudyID@greensunmedical.com. More information about the app is provided in the section: Additional Information on Assessments

Visit 2 (1-2 weeks after Baseline, approximately 1 hour)

1. Standing coronal full-spine radiographs in the GSM brace (5 minutes)
2. Completion of GSM App Feedback Questionnaire (optional)
3. Safety Check: Query for adverse events and other issues
4. Performance Check

   1. If the Cobb angle obtained in the GSM brace is less than, or no more than, 10 degrees greater than that measured in the TLSO (measurement from Baseline Visit 1) then the GSM in-brace correction will be considered equivalent to the standard brace, and the subject will be sent home for a 2-week trial of the GSM brace
   2. If the in-brace Cobb angle is >10 degrees than that in the TLSO, the subject will exit the trial and continue with their current TLSO.
5. The subject will be provided with instructions for removal of the first iButton from the GSM brace 2 weeks following their Baseline visit (corresponding to the storage capacity of the sensors) along with mailing labels and envelopes, and GSM brace diaries.

Phone Visit and Performance Check (2 weeks after baseline)

1. Study staff will contact the subject and parent/guardian to see how well the subject is adapting to the GSM brace and remind the subject/parent to remove the temperature monitor from the brace and send by courier overnight to the study site.
2. Safety Check: Query for adverse events and other issues
3. Performance Check - to insure adherence to prescribed number of hours per day in the GSM brace:

1. If any problems are noted during the phone contact the PI will determine whether adjustments to the brace could alleviate the issues and, if so, ask the subject return to clinic 2. If the temperature monitor data indicate the subject is wearing the GSM brace an average of 2 or more hours less per day than prescribed

1. The PI will determine whether adjustments to the brace could alleviate the issues and have the subject return to clinic; if not, the subject will exit the study and return to their current TLSO
2. If after adjustments to the brace, the subject feels that the brace is still incompatible with the prescribed wear time, the subject will exit the study and return to their current TLSO

Phone Visits (Weeks 4, 6, 8, and 10 after baseline)

1. Study staff will contact the subject and parent/guardian to see how well the subject is adapting to the GSM brace and remind the subject to continue filling out and sending in diaries to the study site in prepaid envelopes.
2. Safety Check: Query for adverse events and other issues

Visit 3 (3-4 months after baseline, approximately 1 hour)

1. Standing coronal full-spine radiographs out of the brace and measurement of the Cobb angle
2. Removal of iButton #2 and download of temperature monitor data
3. Collection of GSM Brace Diary
4. Completion of the Brace Questionnaire and the Italian Spine Youth Quality of Life (ISYQOL) questionnaire
5. Completion of GSM App Feedback Questionnaire (optional)
6. Safety Check: Query for adverse events and other issues
7. Performance Check:

   1. If the Cobb angle measures no more than 10 degrees greater than that obtained from the subject's most recent out of brace radiograph (prior to enrollment), we will conclude the curve is stable or has progressed within the expected limit. If not, the subject will resume use of the TLSO.
   2. If curve stabilization is seen, subjects may opt to continue the GSM brace or resume use of their TLSO based on subject and parent preferences.

Ongoing Evaluations after Visit 3 (following the standard-of-care until GSM brace is discontinued) For subjects continuing to use the GSM brace after Visit 3: Subject clinical care and evaluations (x-rays, clinical exams) after Visit 3 will be limited to that typically performed as the standard of care (SOC). The exception to the SOC will be the administration of the BrQ and ISYQOL at the end of treatment, ongoing monitoring and recording of AE's discovered during routine clinic visits or other communications, and temperature monitoring (at sites where this is not typically SOC). Clinical and radiographic data from these visits will be collected for study purposes (height, weight, onset of menses, Cobb angle(s), kyphosis, lordosis, coronal and sagittal balance, apical vertebral rotation, in-brace Cobb angle(s), and skeletal maturity indicators) as available.

GSM brace treatment will be discontinued using individualized SOC parameters such as Cobb angle and skeletal maturity indicators, at which time the subject will exit the study.

Exit From Study Subjects will exit the study upon occurrence of the following events

1. Visit 2. GSM in-brace Cobb is >10° more than the TLSO in-brace Cobb
2. Subject not wearing or tolerating GSM brace (per temperature monitor reading 2 weeks after baseline, or at any time during study period)
3. Visit 3. GSM out-of-brace Cobb indicates curve progression
4. GSM brace is discontinued using standard of care criteria

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIS
* Current treatment with a TLSO, of ≥5 months' duration
* Existing 3D surface scan of torso and out-of-brace x-ray within the past 6 months. If no scan exists, patient must be willing to undergo a scan to allow fabrication of the GSM brace.
* One curve apex below T7
* Female sex (85% of the AIS population is female)
* Ability to read and write English
* Age 10-15 years

Exclusion Criteria:

* Parents/patients who decline participation and/or do not sign the consent/assent documents
* Pregnant women
* Patients who are unwilling or unable to return for follow-up visits
* Patients who are unable to read and write in English.

Ages: 10 Years to 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-07 (Estimated)

PRIMARY OUTCOMES:
Cobb Angle (Visit 2) | Visit 2 (1 week after baseline)
  Visit 2 GSM in-brace Cobb angle compared to that in the TLSO at baseline
Cobb Angle (Visit 3) | Visit 3 (3 months after Baseline)
  2. Visit 3 out of brace Cobb angle compared to measurements from the most recent out of brace radiograph
GSM Brace wear time | Visit 3 (3 months after baseline)
  3. Average hours of GSM brace wear per day over the 3 month trial period (temperature monitor data)
Brace questionnaire | Visit 3 (3 months after baseline)
  Change in scores on the Brace Questionnaire from baseline to the 3 month Visit.
  Brace questionnaire minimum/maximum values: 0-34 min/max values; lower score is defined as positive feeling/outcome of brace wear while higher score shows negative feeling/outcome towards brace.
Italian Spine Youth Quality of Life | Visit 3 (3 months after baseline)
  Change in scores of the Italian Spine Youth Quality of Life (ISYQOL) from baseline to the 3 month Visit.
  ISYQOL minimum/maximum values: 1-10 min/max values; lower value is defined as disliking brace while higher value is defined as "loving" brace.

SECONDARY OUTCOMES:
% Full Vital Capacity Lung Function Test | Visit 1 (baseline)
  Vital capacity relative to that obtained in the TLSO at Visit 1 and compared between the TSLO Rigid brace vs. Green Sun Medical Brace.
  This will be done via pulmonary function test (% relative to standard norms). Full vital capacity (FVC) function test will be done and assessed at the baseline visit.
Range of Motion (flexion, extension, side bend) | Visit 1 (baseline)
  Range of motion testing involves forward bending (flexion), backwards bending (Extension), side bending on both right and left while wearing both the TLSO rigid brace vs. Green Sun Medical brace. Units will be in cm. Measurement will be done from the floor to the tip of the finger as the subject bends over.
Accelerometer data | Visit 3 (3 months after baseline)
  Accelerometer data (obtained from an embedded sensor in the GSM brace) as an estimate of the average hours of wear per day (to be validated by comparison with temperature monitor data)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Illingworth, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No